CLINICAL TRIAL: NCT06665425
Title: An Open-label, Crossover, Phase 1 Clinical Trial to Evaluate the Pharmacokinetic/Pharmacodynamic Drug-drug Interactions and Safety/Tolerability of Epaminurad and C2406 When Co-administered in Healthy Adults
Brief Title: PK,PD and DDI of Epaminurad and C2406 in Healthy Volunteers
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JW24103
Record Dates: First submitted 2024-10-28; First posted 2024-10-30 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2024-10

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Epaminurad 9mg, C2406 0.6mg
  Interventions: Drug: Epaminurad 9 mg; Drug: C2406

INTERVENTIONS:
Drug: Epaminurad 9 mg — Period 1: Epaminurad / Period 2: C2406 -> Epaminurad + C2406
Drug: C2406 — Period 1: Epaminurad / Period 2: C2406 -> Epaminurad + C2406

SUMMARY:
A Phase 1 Study to evaluate the safety, PK/PD, drug-drug interaction(DDI) of Epaminurad and C2406 in Healthy Volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Age: 19~50
2. Weight: between 50.0 kg~90.0 kg, Body Mass Index(BMI): 18.0 kg/m^2 or heavier and below 30.0 kg/m^2

Exclusion Criteria:

1. Medical history- chronic liver disease, acute gout attack, uric acid stone, diabetes, hypertension, hyperlipidemia or lipid abnormality
2. Clinical examination

   * eGFR (CKD-EPI) < 90mL/min/1.73m^2
   * Serum uric acid < 3 mg/dL or > 7 mg/dL
   * AST (SGOT), ALT (SGPT) > upper limit of normal ranges X 1.5
   * Total bilirubin, γ-GTP > upper limit of normal ranges X 1.5
   * CK > upper limit of normal ranges X 2
   * Positive serologic results

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2025-05-02 (Actual); Study Completion 2025-09-07 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | 7 days
  To evaluate the AUC of Epaminurad and C2406
Peak plasma concentrations (Cmax) | 7 days
  To evaluate the Cmax of Epaminurad and C2406

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-sang Yu, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital Clinical Trials Center, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No